CLINICAL TRIAL: NCT03528044
Title: Evaluation and Follow up of Emotional Regulation, Cognition, Impulsivity and Reward System in Obesity, and Determination of Its Biopsychosocial Risk Factors: A Prospective Study of Obese Patients Before and After Bariatric Surgery
Brief Title: Emotional Regulation, Cognition, Impulsivity and Reward System in Obesity: A Prospective Study of Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Fatih Sultan Mehmet Training and Research Hospital (Other); Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KocU Bari; 2017.081.IRB1.011 (Other: Koc University IRB)
Record Dates: First submitted 2018-03-19; First posted 2018-05-17 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Cognitive Disorder
Keywords: Bariatric surgery; Reward; Cognition; Working memory; Grey matter; GLP-1; Inflammation; Stress; Follow-up; Psychiatric
MeSH Terms: conditions — Obesity; Cognitive Dysfunction; Inflammation | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: In this study, patients undergoing bariatric surgery will be assessed at baseline and after bariatric surgery. We intend to analyze the changes in this repeated and dependent measurements. The other group will be undisturbed during the follow up except for clinical assessments and MRI imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing bariatric surgery (Experimental): In this study, patients will undergo sleeve gastrectomy to reduce the size of the stomach to induce weight loss.
  Interventions: Procedure: Bariatric surgery
- Control group (No Intervention): Healthy controls with normal BMI.

INTERVENTIONS:
Procedure: Bariatric surgery — In this study, patients will undergo sleeve gastrectomy to reduce the size of the stomach to induce weight loss.
  Arms: Patients undergoing bariatric surgery

SUMMARY:
This research investigates obesity and associated psychiatric symptoms and disorders in a wide range of perspectives, to demonstrate the effects of obesity on the brain. The 1st aim is to assess the psychiatric symptom profiles in the group of obese patients applying for bariatric surgery and to determine the associated environmental stress factors. While, it is known that eating disorders, mood disorders and psychiatric drugs can cause obesity, obesity can also cause many psychiatric complications such as depression and cognitive disorders. There are no multi-centered studies that are conducted in this respect, and the guidelines on pre-evaluation and follow-up of patients are also lacking. The 2nd aim is to evaluate and monitor cognitive characteristics before and after bariatric surgery in obese patients. Obese people are at increased risk of dementia and are more likely to have cognitive deficits, especially executive function problems, that can affect everyday life. For this reason, obese individuals should be examined and monitored in more detail in terms of their cognitive characteristics and the change of cognitive functions during the weight loss process. The 3rd aim is to examine the relationship between obesity, bariatric surgery and reward processing system. Studies have been limited in determining whether addiction in these people is due to a search of a continuous substance as a cognitive feature or whether it is difficult to terminate it as an impulsive behavior when encountered with a pleasurable substance, even though there is no reward seeking or reward dependence. The 4th aim is the determination of the neuroanatomical and molecular components of cognitive changes observed after bariatric surgery. During the dynamic process following bariatric surgery, a variety of metabolites, chemokines, and microbiota changes may also affect the brain health and cognition. The 5th aim is to determine factors of eating, emotional regulation, reward system, addiction and impulsivity, and other psychopathologies that cause suboptimal weight loss or weight gain after bariatric surgery. Understanding the psychological and neurobiological factors involved in these processes can improve surgical interventions and significantly increase the quality of life for patients.

DETAILED DESCRIPTION:
Aim 1: To assess the psychiatric symptom profiles in the group of obese patient candidates applying for bariatric surgery and to determine the associated environmental stress factors.

Patients will be evaluated with psychosocial scales as part of their pre-surgery assessments. The first psychosocial evaluation of the patients will be performed by a structured clinical interview (SCID) by Dr. Hale Yapici Eser, Dr. Özge Kılıç and then, the participants will be asked to fill in the self-assessment scales and they will be applied some computer based cognitive tests via the assistance of Candan Yasemin Eren.

Scales used to model environmental factors:

1. Sociodemographic Data Form
2. Childhood Trauma Questionnaire
3. Chronic Stress Scale
4. Perceived Stress Scale
5. Distress Thermometer
6. Multidimensional Scale of Perceived Social Support

   Scales used to evaluate psychiatric symptom profile:
7. Beck Depression Scale
8. Beck Anxiety Scale
9. Barratt Impulsivity Scale
10. Cognitive Failures Questionnaire
11. Mood Disorder Questionnaire
12. Yale Food Addiction Scale
13. Relationship Scales Questionnaire
14. Difficulties in Emotion Regulation Scale
15. Snaith-Hamilton Pleasure Scale

Patients will fill these measurements using Qualtrics. The findings of the structured interview and results of the scale scores will be analyzed by SPSS. From these scales, evaluations other than scales 2 and 13 will be re-administered at the 3rd month and 12th months after bariatric surgery. Scale scores will be used for follow-up of patients.

Aim 2: To evaluate and monitor cognitive characteristics before and after bariatric surgery in obese patients.

The cognitive functions of the patients will be assessed, pre and post operationally (3rd and 12th months), by the Penn-CNP neuropsychological test battery and the 'Cognitive Failures Questionnaire' indicated as the 10th item above. 'Cognitive Failures Questionnaire' is a self-administered scale, which is aimed at questioning the different areas of cognition such as attention, memory and perception. Penn-CNP is a neuropsychological test battery developed by Prof. Dr. Rachel Gur at the University of Pennsylvania and already in use on large sampled and multi centered researches. The required tasks of this battery is translated into Turkish by establishing a connection between Dr. Hale Yapici Eser and these research centers.

The Penn-CNP neuropsychological test battery can assess cognitive features such as emotion recognition and discrimination, working memory, visual-spatial perception and memory, motor praxis, impulsivity and attention. Some of these tests are aimed at evaluating the effect of reaction time and motor capacity on test responses, while others investigate emotion recognition processes with different aspects of cognition such as attention, working and long-term memory, executive functions and visual-spatial perception.For each test applied with this battery, the test results are automatically calculated by the system and the response time, correct and incorrect answers for each response are also presented in an analytical data format. The program also does unbiased arithmetic calculations on important data for further analysis.

Test result tables of the battery can be reviewed in detail from the following link:

https://penncnp.med.upenn.edu/doc.pl?section=pi&content=factsheets/penncnp_test_descriptions-v1.00.pdf

Cognitive scales will be repeated at 0, 3 and 12 months post-operation. These follow-ups have important implications. Findings obtained for each test will be monitored in terms of changes between pre and post operation. Also, the effects of the variables mentioned in method 4 will be analyzed on the scores obtained on each cognitive test by the SPSS program. In addition, test results will be compared in terms of the changes made in the measurements in the control group mentioned in method 4.

Aim 3: To examine the relationship between obesity, bariatric surgery and reward processing system.

The cognitive functions of the patients will be assessed with the "Probabilistic Reward Task (PRT)" pre and 3rd and 12th months after bariatric surgery to examine the changes in the reward learning systems after bariatric surgery.PRT is a signal detection task used for measuring hedonic capacity and reward learning based on monetary reward enhancement. Developed by Diego Pizzagalli in 2005, PRT is an objective assessment of the participants' tendency to modulate their behavior in relation to the prize. At each trial, subjects are asked to choose between two very similar stimuli. The stimuli consist of simple cartoon faces presented at the center of the monitor. Subjects are instructed to press on the appropriate button to determine whether the stimulus is presented with long (11 mm) or short (10 mm) mouth. One of the stimuli (the "rich stimulus") is awarded three times more often than the other ("lean") but the subjects do not know about it. The reward is presented with: "True! You have earned 25 cents". In healthy controls, this reinforcement method leads to response bias, and more frequent rewarding stimuli are preferred. The response bias towards the more frequently rewarded stimuli will be used to operationalize reward sensitivity. Due to participation and validity of the test participants will be given 20 TL independently from their performance. Mentioned evaluations will be repeated at 0, 3 and 12 months. Findings obtained for each test will be monitored in terms of changes between pre and post operation. Also, the effects of the variables mentioned in method 4 will be analyzed on the scores obtained on each cognitive test by the SPSS program.

Aim 4: Determination of the neuroanatomical and molecular components of cognitive changes observed after bariatric surgery.

In this part of the study, brain imaging and biochemical measurements will be conducted. Patients who have completed Method 1 will be evaluated on psychiatric examination and scale scores to be able to be eligible for this stage. During the preliminary evaluations, people with conditions that might affect their cognition and cause brain damage will not be included. Patients who meet the criteria will be exposed to the following measurements at pre-operative, 3 and 12 months. A second group of healthy volunteers with normal body mass index, paired with age, gender, education status and psychiatric assessment scale scores, with normal BMI, will be formed.

Imaging studies: Structural and functional changes in the brain will be evaluated by magnetic resonance imaging (MRI). Thin-section T1-weighted images for evaluation of gray matter changes, resting functional magnetic resonance images for evaluation of functional changes will be obtained. For resting fMRI, patients will be asked to rest eyes closed for 6 minutes without thinking anything. MRI examination will be repeated both for the obese patient group and concurrently healthy controls before surgery (0 months) and after surgery at 3 and 12 months. Imaging will take approximately 30 minutes.

All brain group analyzes of the structural imaging data obtained at the pre-operative, baseline, time point of the obese patient group and the healthy control group will be performed and the brain regions in the obese patient group will be determined for the gray matter changes. The first stage analysis will focus on the brain areas where gray matter changes are observed, and these areas will be compared with the data obtained from the after bariatric surgery imaging sessions. For the evaluation of these changes, focus areas will be placed in the brain areas where obese individuals have gray matter changes, and detailed analysis will be made. Focused analysis and whole brain comparisons performed by placing the areas of interest as mentioned will be performed in comparison with longitudinal data (comparing baseline-3 and 12 months of obese individuals with each other) and normal healthy groups' 3 and 12 months data. In addition, structural changes in the brain will be analyzed in relation to cognitive functions, stress factors, and mood changes. For second stage analysis, interest areas will be placed to the prefrontal cortex, hippocampus, and temporal lobe and data of obese patient group and healthy controls will be compared at the baseline, 3rd and 12th months. In addition, a longitudinal analysis will be performed on the obese patient group (comparing 0-3 and 12 months of obese individuals with each other) to assess the effect of bariatric surgery on these brain areas.

In resting state fMRI, the focus now is to examine the functional connectivity changes in the ventral tegmental area as its activity correlates with reward learning and prefrontal cortex as the center for executive functions. Depending on the findings of the clinical data obtained from the study, different areas of interest will be identified and functional associations will be examined. Focused analyzes on areas of interest mentioned above will be performed both longitudinally (comparing 0-3 and 12 months of the obese individuals with each other) and 3 and 12 months comparisons between healthy controls and obese group. In addition, functional changes in the brain will be analyzed in relation to cognitive functions and mood changes.

Biological Analysis: Blood samples obtained will also be used to analyze peripheral biological markers that may be risk factors. Metabolic parameters, inflammatory markers, and GLP levels will be measured and recorded.

1. Serum cortisol levels
2. Serum GLP levels
3. Ghrelin, leptin
4. Calculation of HbA1C, glucose, insulin levels and HOMA IR
5. Thyroid stimulating hormone (TSH) levels
6. CRP levels
7. Inflammatory panel (IL-1, IL-6 and TNF-a levels)
8. B12, folic acid and ferritin levels
9. Serum lipid profile (total cholesterol, LDL cholesterol, HDL cholesterol, triglyceride)
10. Liver function tests

In addition to neuroanatomical and other biomarkers, investigating physicians will monitor the general clinical status of the patients and changes such as hypertension and sleep apnea will be noted. Nutritionists will also follow diet compliance of the patients. Daily mobility and exercise levels will also be assessed. All of these obtained markers will be used both longitudinally (0-3 and 12 months of obese individuals compared to each other) and comparison to healthy controls at the 0, 3 and 12 months. During the collection of imaging and biomarkers data, the control group will be monitored for 12 months as well.

Aim 5: To determine factors of eating, emotional regulation, reward system, addiction and impulsivity, and other psychopathologies that cause suboptimal weight loss or weight gain after bariatric surgery.

Similar to the previous methods, patients will fill in the self-assessment scales and apply cognitive tests on the computer via the assistance of Candan Yasemin Eren. The tests to be applied in this section will be the scales used to evaluate the environmental and psychiatric profile described in method 1, the PENN-CNP battery described in method 2, and the PRT batteries in method 3.

ELIGIBILITY:
For obese patient group:

Inclusion Criteria:

1. Be between the ages of 18-65
2. To be able to give informed consent
3. Be a candidate for bariatric surgery.

Exclusion Criteria:

1. Dementia
2. Individuals with severe mental retardation and marked cognitive impairments
3. Psychotic disorders
4. Psychoactive substance addiction diagnosis

For healthy volunteers:

Inclusion criteria:

1. Be between the ages of 18-65
2. To be able to give informed consent
3. To be in normal range for BMI
4. To be observed as in the normal mental status examination

Exclusion criteria:

1. Dementia
2. Individuals with severe mental retardation and marked cognitive impairments
3. Psychotic disorders
4. Psychoactive substance addiction diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Changes in working memory following bariatric surgery | Pre-surgery, 3rd and 12th months after bariatric surgery
  Letter-and-Back Task in the PENN-CNP neuropsychological battery will be used to assess working memory. Letter-and-Back asks participants to focus on letters on the screen and press the spacebar according to certain rules. The task consists of three parts: 0-back, 1-back, 2-back. During 0-back, participants press the spacebar when they see letter "X" on the screen. During 1-back, participants press the spacebar when they see the same letter twice. During 2-back, participants press the spacebar when the letter on the screen is the same as the letter before the previous letter.
Grey-matter changes in the entire brain, focused assessments on brain areas known to be associated with cognitive functions | MRI examination will be repeated both for the obese patient group and concurrently healthy controls before surgery (0 months) and after surgery at 3 and 12 months.
  Structural and functional changes in the brain will be evaluated by magnetic resonance imaging (MRI). Thin-section T1-weighted images for evaluation of gray matter changes, resting functional magnetic resonance images for evaluation of functional changes will be obtained. For resting fMRI, patients will be asked to rest eyes closed for 6 minutes without thinking anything. Imaging will take approximately 30 minutes.

SECONDARY OUTCOMES:
Changes in impulsivity following bariatric surgery | Pre-surgery, 3rd and 12th months after bariatric surgery
  Continuous performance task in the PENN-CNP neuropsychological battery and Barratt Impulsivity Scale will be used to assess impulsivity. While continuous performance task assess impulsivity by a computer-based task, Baratt Impulsivity measure is a self-report measure. Therefore, both methods are significant in assessment of impulsivity.
Success of surgery | 3rd and 12th months after bariatric surgery
  Percentage of weight loss proportional to baseline weight measurements
Changes in inflammator factors following bariatric surgery | Pre-surgery, 3rd and 12th months after bariatric surgery
  Blood samples will be obtained from patients to analyze inflammatory markers such as IL-1, IL-6 and TNF-a levels.
Changes in GLP1 will be analyzed following bariatric surgery | Pre-surgery, 3rd and 12th months after bariatric surgery
  Blood samples will be obtained from patients to analyze GLP1 levels.
Changes in social cognition following bariatric surgery | Pre-surgery, 3rd and 12th months after bariatric surgery
  Emotion Recognition Task in the PENN-CNP neuropsychological battery will be used to assess social cognition. Participants see series of 40 faces and are asked to determine the emotion the faces are showing in each trial. There are five different choices: happy, sad, anger, fear and no emotion. The scoring is based on the number of correct responses for each emotion and the number of correctly identified mild and intense emotion expressions. Median response times are also calculated.
Changes in reward learning following bariatric surgery | Pre-surgery, 3rd and 12th months after bariatric surgery
  PRT is used to examine the changes in the reward learning systems after bariatric surgery. It is a signal detection task used for measuring hedonic capacity and reward learning based on monetary reward enhancement. PRT is an objective assessment of the participants' tendency to modulate their behavior in relation to the prize.

CONTACTS AND LOCATIONS:
Overall Officials: Hale Yapici Eser, MD, PHD, Principal Investigator — Koc University School of Medicine
Locations (3):
- Turkey (Türkiye) (3):
  - Fatih Sultan Mehmed Training and Research Hospital, Istanbul
  - Koc University School of Medicine, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Admon R, Pizzagalli DA. Dysfunctional Reward Processing in Depression. Curr Opin Psychol. 2015 Aug 1;4:114-118. doi: 10.1016/j.copsyc.2014.12.011. PMID 26258159
- [Background] Alciati A, Gesuele F, Rizzi A, Sarzi-Puttini P, Foschi D. Childhood parental loss and bipolar spectrum in obese bariatric surgery candidates. Int J Psychiatry Med. 2011;41(2):155-71. doi: 10.2190/PM.41.2.e. PMID 21675347
- [Background] Zeki Al Hazzouri A, Haan MN, Whitmer RA, Yaffe K, Neuhaus J. Central obesity, leptin and cognitive decline: the Sacramento Area Latino Study on Aging. Dement Geriatr Cogn Disord. 2012;33(6):400-9. doi: 10.1159/000339957. Epub 2012 Jul 17. PMID 22814127
- [Background] Alosco ML, Spitznagel MB, Strain G, Devlin M, Cohen R, Crosby RD, Mitchell JE, Gunstad J. Improved serum leptin and ghrelin following bariatric surgery predict better postoperative cognitive function. J Clin Neurol. 2015 Jan;11(1):48-56. doi: 10.3988/jcn.2015.11.1.48. Epub 2015 Jan 2. PMID 25628737
- [Background] Alosco ML, Spitznagel MB, Strain G, Devlin M, Cohen R, Paul R, Crosby RD, Mitchell JE, Gunstad J. Improved memory function two years after bariatric surgery. Obesity (Silver Spring). 2014 Jan;22(1):32-8. doi: 10.1002/oby.20494. Epub 2013 Oct 15. PMID 23625587
- [Background] Anstey KJ, Cherbuin N, Budge M, Young J. Body mass index in midlife and late-life as a risk factor for dementia: a meta-analysis of prospective studies. Obes Rev. 2011 May;12(5):e426-37. doi: 10.1111/j.1467-789X.2010.00825.x. Epub 2011 Feb 23. PMID 21348917
- [Background] Bak M, Seibold-Simpson SM, Darling R. The potential for cross-addiction in post-bariatric surgery patients: Considerations for primary care nurse practitioners. J Am Assoc Nurse Pract. 2016 Dec;28(12):675-682. doi: 10.1002/2327-6924.12390. Epub 2016 Jul 11. PMID 27400415
- [Background] Bellinger FP, Madamba SG, Campbell IL, Siggins GR. Reduced long-term potentiation in the dentate gyrus of transgenic mice with cerebral overexpression of interleukin-6. Neurosci Lett. 1995 Sep 29;198(2):95-8. doi: 10.1016/0304-3940(95)11976-4. PMID 8592650
- [Background] Bergmann KL, Cox SJ, Tabone LE. Influence of a rural environment on patient access and outcomes for bariatric surgery. Surg Obes Relat Dis. 2017 Apr;13(4):632-636. doi: 10.1016/j.soard.2016.11.009. Epub 2016 Nov 11. PMID 28159563
- [Background] Biessels GJ, Deary IJ, Ryan CM. Cognition and diabetes: a lifespan perspective. Lancet Neurol. 2008 Feb;7(2):184-90. doi: 10.1016/S1474-4422(08)70021-8. PMID 18207116
- [Background] Bjorntorp P. Do stress reactions cause abdominal obesity and comorbidities? Obes Rev. 2001 May;2(2):73-86. doi: 10.1046/j.1467-789x.2001.00027.x. PMID 12119665
- [Background] Blum K, Bailey J, Gonzalez AM, Oscar-Berman M, Liu Y, Giordano J, Braverman E, Gold M. Neuro-Genetics of Reward Deficiency Syndrome (RDS) as the Root Cause of "Addiction Transfer": A New Phenomenon Common after Bariatric Surgery. J Genet Syndr Gene Ther. 2011 Dec 23;2012(1):S2-001. doi: 10.4172/2157-7412.S2-001. PMID 23483116
- [Background] Bordignon S, Aparicio MJG, Bertoletti J, Trentini CM. Personality characteristics and bariatric surgery outcomes: a systematic review. Trends Psychiatry Psychother. 2017 Apr-Jun;39(2):124-134. doi: 10.1590/2237-6089-2016-0016. Epub 2017 Jun 12. PMID 28614435
- [Background] Cunningham AJ, Murray CA, O'Neill LA, Lynch MA, O'Connor JJ. Interleukin-1 beta (IL-1 beta) and tumour necrosis factor (TNF) inhibit long-term potentiation in the rat dentate gyrus in vitro. Neurosci Lett. 1996 Jan 12;203(1):17-20. doi: 10.1016/0304-3940(95)12252-4. PMID 8742036
- [Background] Debette S, Seshadri S, Beiser A, Au R, Himali JJ, Palumbo C, Wolf PA, DeCarli C. Midlife vascular risk factor exposure accelerates structural brain aging and cognitive decline. Neurology. 2011 Aug 2;77(5):461-8. doi: 10.1212/WNL.0b013e318227b227. PMID 21810696
- [Background] Dinel AL, Andre C, Aubert A, Ferreira G, Laye S, Castanon N. Cognitive and emotional alterations are related to hippocampal inflammation in a mouse model of metabolic syndrome. PLoS One. 2011;6(9):e24325. doi: 10.1371/journal.pone.0024325. Epub 2011 Sep 16. PMID 21949705
- [Background] Dommes, E., & Georgiewa, P. Grey Matter Volume Differences In Obese As Compared to Normal-Weight Individuals: A Voxel-Based Morphometric Study. Archiv Euromedica, 3(2): 11-16, 2013.
- [Background] Duarte-Guerra LS, Coelho BM, Santo MA, Lotufo-Neto F, Wang YP. Morbidity persistence and comorbidity of mood, anxiety, and eating disorders among preoperative bariatric patients. Psychiatry Res. 2017 Nov;257:1-6. doi: 10.1016/j.psychres.2017.07.020. Epub 2017 Jul 10. PMID 28709116
- [Background] Freese KE, Althouse AD, Ramanathan R, Edwards RP, Bovbjerg DH, Linkov F. Presurgery Weight Loss Goals, Depressive Symptoms, and Weight Loss Among Women Undergoing Bariatric Surgery. Bariatr Surg Pract Patient Care. 2017 Jun 1;12(2):67-71. doi: 10.1089/bari.2016.0038. PMID 28660099
- [Background] Funk LM, Grubber JM, McVay MA, Olsen MK, Yancy WS, Voils CI. Patient predictors of weight loss following a behavioral weight management intervention among US Veterans with severe obesity. Eat Weight Disord. 2018 Oct;23(5):587-595. doi: 10.1007/s40519-017-0425-6. Epub 2017 Aug 29. PMID 28853051
- [Background] Gemma C, Bickford PC. Interleukin-1beta and caspase-1: players in the regulation of age-related cognitive dysfunction. Rev Neurosci. 2007;18(2):137-48. doi: 10.1515/revneuro.2007.18.2.137. PMID 17593876
- [Background] Godard J, Baruch P, Grondin S, Lafleur MF. Psychosocial and neurocognitive functioning in unipolar and bipolar depression: a 12-month prospective study. Psychiatry Res. 2012 Mar 30;196(1):145-53. doi: 10.1016/j.psychres.2011.09.013. Epub 2012 Feb 26. PMID 22370154
- [Background] Gunstad J, Strain G, Devlin MJ, Wing R, Cohen RA, Paul RH, Crosby RD, Mitchell JE. Improved memory function 12 weeks after bariatric surgery. Surg Obes Relat Dis. 2011 Jul-Aug;7(4):465-72. doi: 10.1016/j.soard.2010.09.015. Epub 2010 Oct 30. PMID 21145295
- [Background] Gustafson D, Lissner L, Bengtsson C, Bjorkelund C, Skoog I. A 24-year follow-up of body mass index and cerebral atrophy. Neurology. 2004 Nov 23;63(10):1876-81. doi: 10.1212/01.wnl.0000141850.47773.5f. PMID 15557505
- [Background] Hassing LB, Dahl AK, Thorvaldsson V, Berg S, Gatz M, Pedersen NL, Johansson B. Overweight in midlife and risk of dementia: a 40-year follow-up study. Int J Obes (Lond). 2009 Aug;33(8):893-8. doi: 10.1038/ijo.2009.104. Epub 2009 Jun 9. PMID 19506566
- [Background] Hawkins MA, Alosco ML, Spitznagel MB, Strain G, Devlin M, Cohen R, Crosby RD, Mitchell JE, Gunstad J. The Association Between Reduced Inflammation and Cognitive Gains After Bariatric Surgery. Psychosom Med. 2015 Jul-Aug;77(6):688-96. doi: 10.1097/PSY.0000000000000125. PMID 25478707
- [Background] Hensel JM, Grosman Kaplan K, Anvari M, Taylor VH. The impact of history of exposure to abuse on outcomes after bariatric surgery: data from the Ontario Bariatric Registry. Surg Obes Relat Dis. 2016 Sep-Oct;12(8):1441-1446. doi: 10.1016/j.soard.2016.03.016. Epub 2016 Mar 19. PMID 27387698
- [Background] Horstmann A, Fenske WK, Hankir MK. Argument for a non-linear relationship between severity of human obesity and dopaminergic tone. Obes Rev. 2015 Oct;16(10):821-30. doi: 10.1111/obr.12303. Epub 2015 Jun 22. PMID 26098597
- [Background] Hunter RG, Seligsohn M, Rubin TG, Griffiths BB, Ozdemir Y, Pfaff DW, Datson NA, McEwen BS. Stress and corticosteroids regulate rat hippocampal mitochondrial DNA gene expression via the glucocorticoid receptor. Proc Natl Acad Sci U S A. 2016 Aug 9;113(32):9099-104. doi: 10.1073/pnas.1602185113. Epub 2016 Jul 25. PMID 27457949
- [Background] Ionut V, Bergman RN. Mechanisms responsible for excess weight loss after bariatric surgery. J Diabetes Sci Technol. 2011 Sep 1;5(5):1263-82. doi: 10.1177/193229681100500536. PMID 22027328
- [Background] Ivezaj V, Stoeckel LE, Avena NM, Benoit SC, Conason A, Davis JF, Gearhardt AN, Goldman R, Mitchell JE, Ochner CN, Saules KK, Steffen KJ, Stice E, Sogg S. Obesity and addiction: can a complication of surgery help us understand the connection? Obes Rev. 2017 Jul;18(7):765-775. doi: 10.1111/obr.12542. Epub 2017 Apr 21. PMID 28429582
- [Background] Jacques D, Reynaert C, Zdanowicz N. Liaison psychiatry and bariatric surgery: double standards. What are the possibilities for the systematization of the pre-operative psychiatric assessment in Belgium? Psychiatr Danub. 2016 Sep;28(Suppl-1):121-124. PMID 27663821
- [Background] Jeon BT, Jeong EA, Shin HJ, Lee Y, Lee DH, Kim HJ, Kang SS, Cho GJ, Choi WS, Roh GS. Resveratrol attenuates obesity-associated peripheral and central inflammation and improves memory deficit in mice fed a high-fat diet. Diabetes. 2012 Jun;61(6):1444-54. doi: 10.2337/db11-1498. Epub 2012 Feb 23. PMID 22362175
- [Background] Kalarchian MA, Marcus MD, Levine MD, Courcoulas AP, Pilkonis PA, Ringham RM, Soulakova JN, Weissfeld LA, Rofey DL. Psychiatric disorders among bariatric surgery candidates: relationship to obesity and functional health status. Am J Psychiatry. 2007 Feb;164(2):328-34; quiz 374. doi: 10.1176/ajp.2007.164.2.328. PMID 17267797
- [Background] Kalinowski P, Paluszkiewicz R, Wroblewski T, Remiszewski P, Grodzicki M, Bartoszewicz Z, Krawczyk M. Ghrelin, leptin, and glycemic control after sleeve gastrectomy versus Roux-en-Y gastric bypass-results of a randomized clinical trial. Surg Obes Relat Dis. 2017 Feb;13(2):181-188. doi: 10.1016/j.soard.2016.08.025. Epub 2016 Aug 18. PMID 27692906
- [Background] Karlsson HK, Tuulari JJ, Tuominen L, Hirvonen J, Honka H, Parkkola R, Helin S, Salminen P, Nuutila P, Nummenmaa L. Weight loss after bariatric surgery normalizes brain opioid receptors in morbid obesity. Mol Psychiatry. 2016 Aug;21(8):1057-62. doi: 10.1038/mp.2015.153. Epub 2015 Oct 13. PMID 26460230
- [Background] Kim JH, Choi JH. Pathophysiology and clinical characteristics of hypothalamic obesity in children and adolescents. Ann Pediatr Endocrinol Metab. 2013 Dec;18(4):161-7. doi: 10.6065/apem.2013.18.4.161. Epub 2013 Dec 31. PMID 24904871
- [Background] King WC, Chen JY, Courcoulas AP, Dakin GF, Engel SG, Flum DR, Hinojosa MW, Kalarchian MA, Mattar SG, Mitchell JE, Pomp A, Pories WJ, Steffen KJ, White GE, Wolfe BM, Yanovski SZ. Alcohol and other substance use after bariatric surgery: prospective evidence from a U.S. multicenter cohort study. Surg Obes Relat Dis. 2017 Aug;13(8):1392-1402. doi: 10.1016/j.soard.2017.03.021. Epub 2017 Mar 31. PMID 28528115
- [Background] Kodama K, Noda S, Murakami A, Azuma Y, Takeda N, Yamanouchi N, Okada S, Komatsu N, Sato T, Miyazawa Y, Kawamura I. Depressive disorders as psychiatric complications after obesity surgery. Psychiatry Clin Neurosci. 1998 Oct;52(5):471-6. doi: 10.1046/j.1440-1819.1998.00447.x. PMID 10215007
- [Background] Koyama A, O'Brien J, Weuve J, Blacker D, Metti AL, Yaffe K. The role of peripheral inflammatory markers in dementia and Alzheimer's disease: a meta-analysis. J Gerontol A Biol Sci Med Sci. 2013 Apr;68(4):433-40. doi: 10.1093/gerona/gls187. Epub 2012 Sep 14. PMID 22982688
- [Background] Levin RL, Heller W, Mohanty A, Herrington JD, Miller GA. Cognitive deficits in depression and functional specificity of regional brain activity. Cognitive Therapy and Research. 31:211- 233, 2007.
- [Background] Loane DJ, Byrnes KR. Role of microglia in neurotrauma. Neurotherapeutics. 2010 Oct;7(4):366-77. doi: 10.1016/j.nurt.2010.07.002. PMID 20880501
- [Background] Luppino FS, de Wit LM, Bouvy PF, Stijnen T, Cuijpers P, Penninx BW, Zitman FG. Overweight, obesity, and depression: a systematic review and meta-analysis of longitudinal studies. Arch Gen Psychiatry. 2010 Mar;67(3):220-9. doi: 10.1001/archgenpsychiatry.2010.2. PMID 20194822
- [Background] Magdaleno R Jr, Chaim EA, Pareja JC, Turato ER. The psychology of bariatric patient: what replaces obesity? A qualitative research with Brazilian women. Obes Surg. 2011 Mar;21(3):336-9. doi: 10.1007/s11695-009-9824-8. Epub 2009 Mar 21. PMID 19306052
- [Background] Mahony D. Psychological assessments of bariatric surgery patients. Development, reliability, and exploratory factor analysis of the PsyBari. Obes Surg. 2011 Sep;21(9):1395-406. doi: 10.1007/s11695-010-0108-0. PMID 20306154
- [Background] Malik S, Mitchell JE, Engel S, Crosby R, Wonderlich S. Psychopathology in bariatric surgery candidates: a review of studies using structured diagnostic interviews. Compr Psychiatry. 2014 Feb;55(2):248-59. doi: 10.1016/j.comppsych.2013.08.021. Epub 2013 Oct 24. PMID 24290079
- [Background] Marek RJ, Ben-Porath YS, Heinberg LJ. Understanding the role of psychopathology in bariatric surgery outcomes. Obes Rev. 2016 Feb;17(2):126-41. doi: 10.1111/obr.12356. PMID 26783067
- [Background] McIntyre RS, Cha DS, Soczynska JK, Woldeyohannes HO, Gallaugher LA, Kudlow P, Alsuwaidan M, Baskaran A. Cognitive deficits and functional outcomes in major depressive disorder: determinants, substrates, and treatment interventions. Depress Anxiety. 2013 Jun;30(6):515-27. doi: 10.1002/da.22063. Epub 2013 Mar 6. PMID 23468126
- [Background] McLennan SN, Mathias JL. The depression-executive dysfunction (DED) syndrome and response to antidepressants: a meta-analytic review. Int J Geriatr Psychiatry. 2010 Oct;25(10):933-44. doi: 10.1002/gps.2431. PMID 20872927
- [Background] Montesi L, El Ghoch M, Brodosi L, Calugi S, Marchesini G, Dalle Grave R. Long-term weight loss maintenance for obesity: a multidisciplinary approach. Diabetes Metab Syndr Obes. 2016 Feb 26;9:37-46. doi: 10.2147/DMSO.S89836. eCollection 2016. PMID 27013897
- [Background] Norris L. Psychiatric issues in bariatric surgery. Psychiatr Clin North Am. 2007 Dec;30(4):717-38. doi: 10.1016/j.psc.2007.07.011. PMID 17938042
- [Background] Ogden CL, Yanovski SZ, Carroll MD, Flegal KM. The epidemiology of obesity. Gastroenterology. 2007 May;132(6):2087-102. doi: 10.1053/j.gastro.2007.03.052. PMID 17498505
- [Background] Ouchi N, Parker JL, Lugus JJ, Walsh K. Adipokines in inflammation and metabolic disease. Nat Rev Immunol. 2011 Feb;11(2):85-97. doi: 10.1038/nri2921. Epub 2011 Jan 21. PMID 21252989
- [Background] Paul L, van der Heiden C, Hoek HW. Cognitive behavioral therapy and predictors of weight loss in bariatric surgery patients. Curr Opin Psychiatry. 2017 Nov;30(6):474-479. doi: 10.1097/YCO.0000000000000359. PMID 28795980
- [Background] Pohl J, Woodside B, Luheshi GN. Changes in hypothalamically mediated acute-phase inflammatory responses to lipopolysaccharide in diet-induced obese rats. Endocrinology. 2009 Nov;150(11):4901-10. doi: 10.1210/en.2009-0526. Epub 2009 Sep 24. PMID 19797120
- [Background] Prickett C, Brennan L, Stolwyk R. Examining the relationship between obesity and cognitive function: a systematic literature review. Obes Res Clin Pract. 2015 Mar-Apr;9(2):93-113. doi: 10.1016/j.orcp.2014.05.001. Epub 2014 Jun 18. PMID 25890426
- [Background] Rapp SR, Luchsinger JA, Baker LD, Blackburn GL, Hazuda HP, Demos-McDermott KE, Jeffery RW, Keller JN, McCaffery JM, Pajewski NM, Evans M, Wadden TA, Arnold SE, Espeland MA; Look AHEAD Research Group. Effect of a Long-Term Intensive Lifestyle Intervention on Cognitive Function: Action for Health in Diabetes Study. J Am Geriatr Soc. 2017 May;65(5):966-972. doi: 10.1111/jgs.14692. Epub 2017 Jan 9. PMID 28067945
- [Background] Reslan S, Saules KK, Greenwald MK, Schuh LM. Substance misuse following Roux-en-Y gastric bypass surgery. Subst Use Misuse. 2014 Mar;49(4):405-17. doi: 10.3109/10826084.2013.841249. Epub 2013 Oct 8. PMID 24102253
- [Background] Salcedo I, Tweedie D, Li Y, Greig NH. Neuroprotective and neurotrophic actions of glucagon-like peptide-1: an emerging opportunity to treat neurodegenerative and cerebrovascular disorders. Br J Pharmacol. 2012 Jul;166(5):1586-99. doi: 10.1111/j.1476-5381.2012.01971.x. PMID 22519295
- [Background] Schmitt A, Falkai P. Negative symptoms and therapy strategies in schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2015 Oct;265(7):541-2. doi: 10.1007/s00406-015-0637-6. No abstract available. PMID 26319528
- [Background] Scholtz S, Goldstone AP, le Roux CW. Changes in Reward after Gastric Bypass: the Advantages and Disadvantages. Curr Atheroscler Rep. 2015 Oct;17(10):61. doi: 10.1007/s11883-015-0534-5. PMID 26358733
- [Background] Scholtz S, Miras AD, Chhina N, Prechtl CG, Sleeth ML, Daud NM, Ismail NA, Durighel G, Ahmed AR, Olbers T, Vincent RP, Alaghband-Zadeh J, Ghatei MA, Waldman AD, Frost GS, Bell JD, le Roux CW, Goldstone AP. Obese patients after gastric bypass surgery have lower brain-hedonic responses to food than after gastric banding. Gut. 2014 Jun;63(6):891-902. doi: 10.1136/gutjnl-2013-305008. Epub 2013 Aug 20. PMID 23964100
- [Background] Sevincer GM, Konuk N, Bozkurt S, Coskun H. Food addiction and the outcome of bariatric surgery at 1-year: Prospective observational study. Psychiatry Res. 2016 Oct 30;244:159-64. doi: 10.1016/j.psychres.2016.07.022. Epub 2016 Jul 12. PMID 27479107
- [Background] Sockalingam S, Hawa R, Wnuk S, Santiago V, Kowgier M, Jackson T, Okrainec A, Cassin S. Psychosocial predictors of quality of life and weight loss two years after bariatric surgery: Results from the Toronto Bari-PSYCH study. Gen Hosp Psychiatry. 2017 Jul;47:7-13. doi: 10.1016/j.genhosppsych.2017.04.005. Epub 2017 Apr 20. PMID 28807141
- [Background] Spitznagel MB, Hawkins M, Alosco M, Galioto R, Garcia S, Miller L, Gunstad J. Neurocognitive Effects of Obesity and Bariatric Surgery. Eur Eat Disord Rev. 2015 Nov;23(6):488-95. doi: 10.1002/erv.2393. Epub 2015 Aug 19. PMID 26289991
- [Background] Strazzullo P, D'Elia L, Cairella G, Garbagnati F, Cappuccio FP, Scalfi L. Excess body weight and incidence of stroke: meta-analysis of prospective studies with 2 million participants. Stroke. 2010 May;41(5):e418-26. doi: 10.1161/STROKEAHA.109.576967. Epub 2010 Mar 18. PMID 20299666
- [Background] Sturm R. Increases in morbid obesity in the USA: 2000-2005. Public Health. 2007 Jul;121(7):492-6. doi: 10.1016/j.puhe.2007.01.006. Epub 2007 Mar 30. PMID 17399752
- [Background] Terra X, Auguet T, Guiu-Jurado E, Berlanga A, Orellana-Gavalda JM, Hernandez M, Sabench F, Porras JA, Llutart J, Martinez S, Aguilar C, Del Castillo D, Richart C. Long-term changes in leptin, chemerin and ghrelin levels following different bariatric surgery procedures: Roux-en-Y gastric bypass and sleeve gastrectomy. Obes Surg. 2013 Nov;23(11):1790-8. doi: 10.1007/s11695-013-1033-9. PMID 23832521
- [Background] Thiara G, Yanofksy R, Abdul-Kader S, Santiago VA, Cassin S, Okrainec A, Jackson T, Hawa R, Sockalingam S. Toronto Bariatric Interprofessional Psychosocial Assessment Suitability Scale: Evaluating A New Clinical Assessment Tool for Bariatric Surgery Candidates. Psychosomatics. 2016 Mar-Apr;57(2):165-73. doi: 10.1016/j.psym.2015.12.003. Epub 2015 Dec 5. PMID 26895728
- [Background] Thiara G, Cigliobianco M, Muravsky A, Paoli RA, Mansur R, Hawa R, McIntyre RS, Sockalingam S. Evidence for Neurocognitive Improvement After Bariatric Surgery: A Systematic Review. Psychosomatics. 2017 May-Jun;58(3):217-227. doi: 10.1016/j.psym.2017.02.004. Epub 2017 Feb 21. PMID 28410777
- [Background] Titova OE, Hjorth OC, Schioth HB, Brooks SJ. Anorexia nervosa is linked to reduced brain structure in reward and somatosensory regions: a meta-analysis of VBM studies. BMC Psychiatry. 2013 Apr 9;13:110. doi: 10.1186/1471-244X-13-110. PMID 23570420
- [Background] Torres SJ, Nowson CA. Relationship between stress, eating behavior, and obesity. Nutrition. 2007 Nov-Dec;23(11-12):887-94. doi: 10.1016/j.nut.2007.08.008. Epub 2007 Sep 17. PMID 17869482
- [Background] Trivedi MH, Greer TL. Cognitive dysfunction in unipolar depression: implications for treatment. J Affect Disord. 2014 Jan;152-154:19-27. doi: 10.1016/j.jad.2013.09.012. Epub 2013 Sep 25. PMID 24215896
- [Background] Trollor JN, Smith E, Agars E, Kuan SA, Baune BT, Campbell L, Samaras K, Crawford J, Lux O, Kochan NA, Brodaty H, Sachdev P. The association between systemic inflammation and cognitive performance in the elderly: the Sydney Memory and Ageing Study. Age (Dordr). 2012 Oct;34(5):1295-308. doi: 10.1007/s11357-011-9301-x. Epub 2011 Aug 19. PMID 21853262
- [Background] van den Berg E, Kloppenborg RP, Kessels RP, Kappelle LJ, Biessels GJ. Type 2 diabetes mellitus, hypertension, dyslipidemia and obesity: A systematic comparison of their impact on cognition. Biochim Biophys Acta. 2009 May;1792(5):470-81. doi: 10.1016/j.bbadis.2008.09.004. Epub 2008 Sep 23. PMID 18848880
- [Background] Veit R, Kullmann S, Heni M, Machann J, Haring HU, Fritsche A, Preissl H. Reduced cortical thickness associated with visceral fat and BMI. Neuroimage Clin. 2014 Sep 26;6:307-11. doi: 10.1016/j.nicl.2014.09.013. eCollection 2014. PMID 25379443
- [Background] Veronese N, Facchini S, Stubbs B, Luchini C, Solmi M, Manzato E, Sergi G, Maggi S, Cosco T, Fontana L. Weight loss is associated with improvements in cognitive function among overweight and obese people: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2017 Jan;72:87-94. doi: 10.1016/j.neubiorev.2016.11.017. Epub 2016 Nov 24. PMID 27890688
- [Background] Vezzani A, Viviani B. Neuromodulatory properties of inflammatory cytokines and their impact on neuronal excitability. Neuropharmacology. 2015 Sep;96(Pt A):70-82. doi: 10.1016/j.neuropharm.2014.10.027. Epub 2014 Nov 8. PMID 25445483
- [Background] Volkow ND, Wang GJ, Telang F, Fowler JS, Goldstein RZ, Alia-Klein N, Logan J, Wong C, Thanos PK, Ma Y, Pradhan K. Inverse association between BMI and prefrontal metabolic activity in healthy adults. Obesity (Silver Spring). 2009 Jan;17(1):60-5. doi: 10.1038/oby.2008.469. Epub 2008 Oct 23. PMID 18948965
- [Background] Votruba K, Marshall D, Finks J, Giordani B. Neuropsychological factors and bariatric surgery: a review. Curr Psychiatry Rep. 2014 Jun;16(6):448. doi: 10.1007/s11920-014-0448-x. PMID 24740234
- [Background] Wadden TA, Sarwer DB, Fabricatore AN, Jones L, Stack R, Williams NS. Psychosocial and behavioral status of patients undergoing bariatric surgery: what to expect before and after surgery. Med Clin North Am. 2007 May;91(3):451-69, xi-xii. doi: 10.1016/j.mcna.2007.01.003. PMID 17509389
- [Background] Whitmer RA, Gunderson EP, Barrett-Connor E, Quesenberry CP Jr, Yaffe K. Obesity in middle age and future risk of dementia: a 27 year longitudinal population based study. BMJ. 2005 Jun 11;330(7504):1360. doi: 10.1136/bmj.38446.466238.E0. Epub 2005 Apr 29. PMID 15863436
- [Background] Yirmiya R, Goshen I. Immune modulation of learning, memory, neural plasticity and neurogenesis. Brain Behav Immun. 2011 Feb;25(2):181-213. doi: 10.1016/j.bbi.2010.10.015. Epub 2010 Oct 21. PMID 20970492
- [Background] Zhang Y, Ji G, Xu M, Cai W, Zhu Q, Qian L, Zhang YE, Yuan K, Liu J, Li Q, Cui G, Wang H, Zhao Q, Wu K, Fan D, Gold MS, Tian J, Tomasi D, Liu Y, Nie Y, Wang GJ. Recovery of brain structural abnormalities in morbidly obese patients after bariatric surgery. Int J Obes (Lond). 2016 Oct;40(10):1558-1565. doi: 10.1038/ijo.2016.98. Epub 2016 May 20. PMID 27200505
- [Background] Zimmerman M, Francione-Witt C, Chelminski I, Young D, Boerescu D, Attiullah N, Pohl D, Roye GD, Harrington DT. Presurgical psychiatric evaluations of candidates for bariatric surgery, part 1: reliability and reasons for and frequency of exclusion. J Clin Psychiatry. 2007 Oct;68(10):1557-62. doi: 10.4088/jcp.v68n1014. PMID 17960972